CLINICAL TRIAL: NCT05336838
Title: Use of Quantra® System in Clinical Practice to Improve Management of Post-partum Haemorrhage : a Prospective Study
Brief Title: Improving Management of Post-partum Haemorrhage With Quantra® System
Acronym: Quantralab
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Principal Investigator, GRENIE, Doctor, University Hospital, Montpellier
Other Study IDs: RECHMPL21_0729
Record Dates: First submitted 2022-03-23; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Post Partum Haemorrhage
Keywords: Post partum haemorrhage; Bleeding; Labour; Vaginal delivery; Caesarean section
MeSH Terms: conditions — Postpartum Hemorrhage; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post partum haemorrhage is a concerning situation in maternity wards, though it is not the first cause of maternal mortality anymore.

It has been already shown that low fibrinogen level is a major predictive factor of massive bleeding after delivery.

In this situation, the early knowledge of fibrinogen level could enhance care of women experiencing post partum haemorrhage.

In a cohort of women suffering from post partum haemorrhage, this study will evaluate whether assessing fibrinogen level would be faster using the Quantra® system than the standard coagulation test.

ELIGIBILITY:
Inclusion Criteria:

Women ≥ 18 years old Experiencing post partum haemorrhage ≥ 500 mL Within 24 hours after delivery

Exclusion Criteria:

* Previous anemia ≤ 7g/dL
* Known bleeding disorders
* Ongoing antiplatelets treatment
* Ongoing anticoagulant treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women ≥ 18 years old experiencing post partum haemorrhage ≥ 500 mL
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of delay in obtaining Quantra Fibrinogen Clot Stiffness result to standard fibrinogen level result | When post partum haemorrhage occurred, within 24 hours after delivery
  Comparison of delay in obtaining Quantra Fibrinogen Clot Stiffness result to standard fibrinogen level result

SECONDARY OUTCOMES:
Comparison of level of fibrinogen assessed by Quantra Fibrinogen Clot Stiffness to level of fibrinogen assessed by standard coagulation test | When post partum haemorrhage occurred, within 24 hours after delivery
  Fibrinogen level assessed by Quantra and standard coagulation tests
Comparison of Quantra Clot Time result to Standard Kaolin Clotting time result | When post partum haemorrhage occurred, within 24 hours after delivery
  Coagulation function assessed by Quantra and standard coagulation tests
Comparison of Platelet Clot Stiffness result to standard platelet count result | When post partum haemorrhage occurred, within 24 hours after delivery
  Platelet function assessed by Quantra and standard platelet count.
Rate of satisfaction of anesthetist in charge of patient assessed by Lickert scale | When post partum haemorrhage occurred, within 24 hours after delivery
  Rate of satisfaction of anesthetist in charge of patient assessed by Lickert scale [1-Strongly disagree ; 2-Disagree ; 3-Neither agree nor disagree ; 4-Agree ; 5-Strongly agree